CLINICAL TRIAL: NCT07064304
Title: Clinical Efficacy of Er,Cr:YSGG Laser for Deepithelialization of Free Gingival Grafts in Gingival Recession Treatment: A Randomized, Split-Mouth Clinical Trial
Brief Title: Er,Cr:YSGG Laser for Deepithelialization in Gingival Recession.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: WroclawMU6
Record Dates: First submitted 2025-06-30; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Gingival Recession, Localized; Keratinized Tissue; Gingival Thickness; Pocket Depth
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Deepithelialization (LDEE) (Experimental): In this arm, deepithelialization of the free gingival graft was performed extraorally using an Er,Cr:YSGG laser (2780 nm; 2.5 W; 83.3 mJ; 30 Hz; 600 μm tip) before graft placement at the recipient site.
  Interventions: Procedure: Laser Deepithelialization of Free Gingival Graft
- Scalpel Deepithelialization (DEE) (Active Comparator): In this arm, the epithelium was removed manually using a 15c surgical scalpel from the harvested palatal free gingival graft before placement.
  Interventions: Procedure: Scalpel Deepithelialization of Free Gingival Graft

INTERVENTIONS:
Procedure: Laser Deepithelialization of Free Gingival Graft — Extraoral deepithelialization of harvested free gingival graft using Er,Cr:YSGG laser (2780 nm, 2.5 W, 83.3 mJ, 30 Hz, 600 μm tip) before placement in gingival recession treatment.
  Arms: Laser Deepithelialization (LDEE)
Procedure: Scalpel Deepithelialization of Free Gingival Graft — Extraoral deepithelialization of harvested free gingival graft using a 15c surgical scalpel blade before placement in gingival recession treatment.
  Arms: Scalpel Deepithelialization (DEE)

SUMMARY:
Abstract: Introduction: The deepithelialized free gingival graft (DGG) technique provides high-quality connective tissue grafts (CTGs) with predictable outcomes for recession cov-erage. This study evaluates a novel method of free gingival graft (FGG) deepithelialization using an Er,Cr:YSGG laser (LDEE) for treating multiple gingival recessions. Methods: A split-mouth study was conducted on 46 (n=46) recessions in 9 patients (23 per test and control group). Sites were randomized. Full-thickness palatal grafts were harvested with a scalpel. In the test group (LDEE), deepithelialization was performed extraorally using an Er,Cr:YSGG laser (2780 nm; 2.5 W, 83.3 mJ, 30 Hz, 600 µm tip). In the control group (DEE), a 15c scalpel was used. All CTGs were applied using the modified coronally advanced tunnel (TUN) technique. Clinical parameters-recession depth (RD), keratinized tissue width (KT), gingival thickness (GT), pocket depth (PD), clinical attachment loss (CAL), pink esthetic score (PES), approximal plaque index (API), mean root coverage (MRC), and complete root coverage (CRC)-were assessed at baseline (T0), 3 months (T1), and 6 months (T2). Results: Both LDEE and DEE groups showed significant improvements in RD, KT, GT, PD, and CAL over time (p < 0.001). At T1 and T2, KT was significantly higher in the LDEE group (T1: 3.73±0.72 mm; T2: 3.98±0.76 mm) compared to the DEE group (T1: 3.21±0.61 mm; T2: 3.44±0.74 mm; p < 0.05). Other parameters (RD, GT, PD, CAL) showed no statistically significant intergroup differences at any time point (p > 0.05). After 6 months, MRC was 95% and CRC 82.6% for LDEE, compared to 94.8% and 82.6% for DEE (p > 0.05). PES scores were similar between groups at all time points (p > 0.05). Conclusion: Both laser- and scalpel-deepithelialized grafts effectively treated gingival recessions. LDEE combined with TUN resulted in significantly greater KT width compared to DEE + TUN.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Presence of multiple Miller Class I or II gingival recessions
* Good general and oral health
* Patient consent to participate in the clinical trial
* Availability for follow-up at 3 and 6 months

Exclusion Criteria:

* Smoking or history of smoking in the last 6 months
* Systemic diseases affecting wound healing (e.g., diabetes, immunodeficiencies)
* Pregnancy or lactation
* Use of medications that influence periodontal tissues (e.g., immunosuppressants, corticosteroids)
* History of periodontal surgery in the area of interest within the past 12 months Inadequate oral hygiene (plaque index >20%)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Recession Depth | Baseline, 3 months, and 6 months postoperatively
  Measurement of gingival recession depth in millimeters to evaluate soft tissue response to treatment.
  Unit of Measure: mm
Change in Keratinized Tissue Width | Baseline, 3 months, and 6 months postoperatively
  Measurement of the width of keratinized gingiva in millimeters from the mucogingival junction to the free gingival margin.
  Unit of Measure: mm
Change in Gingival Thickness | Baseline, 3 months, and 6 months postoperatively
  Assessment of gingival tissue thickness using a standardized probe. Unit of Measure: mm
Change in Pocket Depth | Baseline, 3 months, and 6 months postoperatively
  Probing depth measured from the gingival margin to the base of the periodontal pocket.
  Unit of Measure: mm
Change in Clinical Attachment Level | Baseline, 3 months, and 6 months postoperatively
  Measurement of the distance from the cementoenamel junction to the base of the periodontal pocket.
  Unit of Measure: mm
Change in Pink Esthetic Score | Baseline, 3 months, and 6 months postoperatively
  Percentage of interdental spaces with visible plaque, calculated to assess oral hygiene status. A lower percentage indicates better plaque control.
  Unit of Measure: percentage (%)
Mean Root Coverage | 6 months postoperatively
  Average percentage of root surface covered by soft tissue following treatment, calculated across all treated sites.
  Unit of Measure: percentage (%)
Complete Root Coverage | 6 months postoperatively
  Proportion of treated sites that achieved 100% root coverage postoperatively. Unit of Measure: percentage (%)

SECONDARY OUTCOMES:
Histopathological Evaluation of Laser-Treated Connective Tissue Grafts | Immediately postoperatively
  Microscopic assessment of grafts treated with Er,Cr:YSGG laser to evaluate the quality of deepithelialization and potential thermal damage. Parameters included the presence of a clear boundary between epithelium and connective tissue, absence of carbonization or necrosis, and preservation of tissue architecture.

CONTACTS AND LOCATIONS:
Locations (1):
- Dentoplex, Bielsko-Biala, Poland

IPD SHARING:
Plan to Share IPD: No
Although this was a prospective clinical study, we do not plan to share individual participant data (IPD) due to lack of consent for data sharing obtained at the time of enrollment.